CLINICAL TRIAL: NCT00276549
Title: Phase II Trial of Gemcitabine And Docetaxel In Androgen-Independent Metastatic Prostate Cancer
Brief Title: Gemcitabine and Docetaxel in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCF7143; P30CA043703 (NIH); CASE-CCF-7143 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Results first posted 2012-06-06 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine and Docetaxel i (Experimental)
  Interventions: Drug: docetaxel; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: docetaxel — docetaxel IV over 60 minutes on day 8. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.
Drug: gemcitabine hydrochloride — IV over 30 minutes on days 1 and 8 followed by docetaxel IV over 60 minutes on day 8. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with docetaxel works in treating patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate and toxicity in patients with androgen-independent metastatic prostate cancer treated with gemcitabine hydrochloride and docetaxel.

OUTLINE: This is an open-label study.

Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8 followed by docetaxel IV over 60 minutes on day 8. Treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for at least 5 years.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Androgen-independent metastatic prostate cancer with evidence of clinical, radiographic, or biochemical progression in the setting of castrate levels of testosterone (< 50 mg/dL)

    * No androgen-independent prostate cancer with a rising prostate-specific antigen (PSA) without clinical or radiographic evidence of metastases
  * Clinical or radiographic evidence of metastatic disease with a rising PSA measured 2 times at ≥ 1 week interval allowed
* Antiandrogen therapy must have been stopped at least 4 weeks (for flutamide) or 6 weeks (for bicalutamide or nilutamide) prior to study entry with evidence of either a rising PSA (from baseline) measured twice at least 2 weeks apart or radiographic evidence of disease progression
* Testicular androgen suppression (< 50 mg/dL) must be maintained with either luteinizing-hormone releasing-hormone (LHRH) therapy or bilateral orchiectomy
* No clinical evidence of CNS metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2 times normal
* Creatinine < 2 mg/dL
* No history of severe uncontrolled congestive heart failure (CHF), ventricular dysrhythmias, or severe cardiovascular disease (American Heart Association class III or IV)
* Disease-free of prior malignancies for ≥ 5 years, with the exception of curatively treated basal cell or squamous cell carcinoma of the skin or low-grade, low-stage bladder cancer
* No active infection or parenteral antibiotics within 7 days of study entry
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No radiation therapy within 4 weeks prior to study entry
* No filgrastim (G-CSF) within 24 hours before or after study therapy
* No prior systemic chemotherapy for metastatic disease

  * Neoadjuvant or adjuvant non-taxane chemotherapy more than 1 year prior to study entry allowed
* No concurrent local radiotherapy for control of pain or life-threatening situations

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dreicer, MD, FACP, Study Chair — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from July 2004-October 2006 from medical clinic.
Groups:
- Gemcitabine (Gemzar) and Docetaxel (Taxotere): Gemcitabine (Gemzar) 800 mg/m2 administered intravenously over 30 to 60 minutes on Day 1 and 8 of each treatment cycle and docetaxel (Taxotere) 75 mg/m2 administered intravenously over 30 to 60 minutes on Day 8 followed the Day 8 infusion of gemcitabine.
Period: Overall Study
Arm/Group | Gemcitabine (Gemzar) and Docetaxel (Taxotere)
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine (Gemzar) and Docetaxel (Taxotere)
Number analyzed (Participants) | 35
Age Continuous [Median (Full Range); unit: years] | 67 [55 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Objective PSA Response Rate (Number of Patients With a PSA Response)
Description: Decline from a baseline value by ≥ 50% or normalization of PSA (< 0.03) confirmed by a second measurement at least 1 week or more weeks later. Patients must not demonstrate clinical or radiographic evidence of disease progression during this time period. The date of response will be defined as the first date at which the PSA declined from baseline by ≥ 50% or normalized.
Time Frame: every 4 weeks
Population: All patients that received treatment.
Measure: Number; unit: participants
Arm/Group | Gemcitabine (Gemzar) and Docetaxel (Taxotere)
Number analyzed (Participants) | 35
participants
  Number of patients with a response ≥ 50% | 17
  Number of patients with no response | 18

2. Primary Outcome: Number of Patients With Measurable Soft Tissue Disease Will be Assessed Per Solid Tumor Response Criteria (RECIST).
Description: Patients who have a response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) by RECIST criteria. To be assigned a status of PR or CR, changes in tumor measurements must be confirmed by repeat assessments that should be performed no less than 4 weeks after the criteria for response are first met. In the case of SD, patients who do not meet the criteria for response or progressive disease for at least 90 days will be categorized as stable disease.
Time Frame: at 4 weeks after treatment completion
Population: 25 patients had RECIST defined measurable disease at study entry. Confirmed response required 2 consecutive measurements at least 1 week later.Three patients did not have follow up measurements therefore were not evaluable.
Measure: Number; unit: participants
Arm/Group | Gemcitabine (Gemzar) and Docetaxel (Taxotere)
Number analyzed (Participants) | 22
participants
  Partial Response | 3
  Stable Disease | 19

ADVERSE EVENTS:
Time Frame: Patients were followed for adverse events while on treatment and on study over a two year time frame.
Arm/Group | Gemcitabine (Gemzar) and Docetaxel (Taxotere)
Serious Adverse Events (participants affected / at risk) | 7/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine (Gemzar) and Docetaxel (Taxotere) (N=35)
Neutropenia (Blood and lymphatic system disorders) | 6
Neutropenia/fever (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine (Gemzar) and Docetaxel (Taxotere) (N=35)
Alopecia (Skin and subcutaneous tissue disorders) | 28
Anemia (Blood and lymphatic system disorders) | 16
Anorexia (Metabolism and nutrition disorders) | 13
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Chills/Rigors (General disorders) | 7
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 10
Dizziness/lightheadedness (Nervous system disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11
Edema (General disorders) | 16
Elevated AST (aspartate aminotransferase); ALT (alanine aminotransferase) (Hepatobiliary disorders) | 7
Fatigue (General disorders) | 28
Fever without Neutropenia (General disorders) | 14
Flushing (Skin and subcutaneous tissue disorders) | 2
Headache/Migraine (Nervous system disorders) | 2
Hot Flashes/Flushes (Endocrine disorders) | 2
Increased Alkaline Phosphatase (Hepatobiliary disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 11
Lymphopenia (Blood and lymphatic system disorders) | 3
Mucositis (oral) (Gastrointestinal disorders) | 6
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2
Myalgia/Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Nail Changes (Skin and subcutaneous tissue disorders) | 6
Nasal Congestion/Drainage (Respiratory, thoracic and mediastinal disorders) | 2
Nausea/vomiting (Gastrointestinal disorders) | 20
Neuropathy (Nervous system disorders) | 9
Neutropenia (Blood and lymphatic system disorders) | 14
Other Gastrointestinal (Gastrointestinal disorders) | 6
Rash/desquamation (Skin and subcutaneous tissue disorders) | 8
Rhinitis (Infections and infestations) | 3
Taste changes (Nervous system disorders) | 15
Tearing (Eye disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Weight Loss (Investigations) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes